CLINICAL TRIAL: NCT02396888
Title: Effects of Local Insulin on Angiogenesis in Acute Wounds in Non-diabetic Patients
Brief Title: Effects of Local Insulin on Wound Angiogenesis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Collaborators: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, MARIO AURELIO MARTÍNEZ-JIMÉNEZ, General Surgeon, Hospital Central "Dr. Ignacio Morones Prieto"
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71-13
Record Dates: First submitted 2015-03-06; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Angiogenesis
Keywords: Blood vessel; Fibroplasia; Wound healing; Insulin
MeSH Terms: conditions — Fibrosis; Insulin Resistance | interventions — Insulin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin (Experimental): Half of the wound surface was treated daily with intermediate insulin. Allocation was randomized.
  Interventions: Drug: Insulin
- Placebo (Placebo Comparator): Half of the wound surface was treated daily with normal saline. Allocation was randomized.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Insulin — Half of the wound surface was treated daily with 10 units of intermediate insulin.
  Arms: Insulin
Drug: Placebo — Half of the wound surface was treated daily with 0.1 cc of normal saline.
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Randomized, split plot, double-blind, placebo controlled trial. Half of the wounds surface was applied daily with insulin and the other half with saline solution as placebo. Biopsy specimens of the two sides were obtained on days 0 and 14. Number of blood vessels will be evaluated as main outcome.

DETAILED DESCRIPTION:
Randomized, split plot, double-blind, placebo controlled trial. Non-diabetic patients with full-thickness wounds will be treated in the following manner: in half of the surface insulin will be applied in a daily basis, on the other half, saline solution will be used as placebo. Biopsy specimens of both sides will be obtained on days 0 and 14. Number of blood vessels will be evaluated as main outcome.

ELIGIBILITY:
Inclusion Criteria:

* Nondiabetic patients with full-thickness acute wounds

Exclusion Criteria:

* Diabetic patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-04 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Number of blood vessels | 14 days
  In a biopsy taken at baseline, blood vessels will be counted

SECONDARY OUTCOMES:
Hypoglycaemia | 14 days
  Presence of capillary blood glucose of <60 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Aguilar-García, MD, Study Chair — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Result] Martinez-Jimenez MA, Aguilar-Garcia J, Valdes-Rodriguez R, Metlich-Medlich MA, Dietsch LJP, Gaitan-Gaona FI, Kolosovas-Machuca ES, Gonzalez FJ, Sanchez-Aguilar JM. Local use of insulin in wounds of diabetic patients: higher temperature, fibrosis, and angiogenesis. Plast Reconstr Surg. 2013 Dec;132(6):1015e-1019e. doi: 10.1097/PRS.0b013e3182a806f0. PMID 24281606